CLINICAL TRIAL: NCT00397033
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Two Dosages of Paliperidone ER in the Treatment of Patients With Schizoaffective Disorder.
Brief Title: Evaluation of Effectiveness and Safety of Paliperidone Extended Release in Patients With Schizoaffective Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR010498; R076477SCA3001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Results first posted 2009-07-28 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Schizoaffective Disorder; Psychotic Disorder
Keywords: Schizoaffective Disorder; antipsychotic; paliperidone; placebo
MeSH Terms: conditions — Psychotic Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 002 (Experimental): Paliperidone ER 12mg/day paliperidone er for 6 weeks
  Interventions: Drug: Paliperidone ER
- 001 (Experimental): Paliperidone ER 6mg/day paliperidone er for 6 weeks
  Interventions: Drug: Paliperidone ER
- 003 (Placebo Comparator): Placebo Placebo for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paliperidone ER — 6mg/day paliperidone er for 6 weeks
  Arms: 001
Drug: Paliperidone ER — 12mg/day paliperidone er for 6 weeks
  Arms: 002
Drug: Placebo — Placebo for 6 weeks
  Arms: 003

SUMMARY:
The purpose of this study is to measure the effectiveness and assess the safety of two dosages of the antipsychotic paliperidone extended-release (ER) in patients who are experiencing an acute episode of schizoaffective disorder.

DETAILED DESCRIPTION:
Schizophrenia and schizoaffective disorder are closely related in terms of symptoms, coexisting conditions, and genetic risk. In previous studies in patients with schizophrenia, treatment with paliperidone extended-release (ER) improved psychotic symptoms, as well as mood symptoms evaluated by anxiety/depression and hostility/excitement Positive and Negative Symptoms of Schizophrenia (PANSS) factor scores. Therefore, paliperidone ER may also be effective in treating symptoms of schizoaffective disorder. Paliperidone's limited potential for drug-drug interaction is particularly important in this patient population, in which multiple drug therapy is relatively common. This multicenter, double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), randomized (patients are assigned different treatments based on chance), placebo-controlled, parallel-group study is designed to examine the effectiveness and safety of paliperidone ER in adult patients with schizoaffective disorder who are experiencing an acute episode of this disorder. Patients in the study will be randomly assigned to 1 of 3 groups to receive 6 weeks of oral treatment with 1 of 2 dosages of paliperidone ER or placebo. The primary efficacy outcome will be the change from baseline to Week 6, or the last post-randomization assessment during double-blind treatment (endpoint), in the PANSS total score. Safety will be assessed by monitoring adverse events, clinical laboratory testing, pregnancy testing, vital signs measurements, physical examination, administration of a 12-lead ECG, movement disorders side effect scales, and the InterSePT Scale for Suicidal Thinking. Patients may also choose to participate in a pharmacogenomic (DNA) analysis. The primary study hypotheses are that at least one of the two dosages of paliperidone ER is better than placebo on the change from baseline in the PANSS total score in acutely ill patients with schizoaffective disorder at the end of 6 weeks of treatment. Patients will receive study drug by mouth for a total of 43 days. Beginning on Day 1, patients will take either placebo or 1 of 2 doses of paliperidone: 6 mg/day (low randomized dosage) or 12 mg/day (high randomized dosage). During the first 2 weeks, dosages may be adjusted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual - Fourth Edition (DSM-IV) diagnosis of schizoaffective disorder
* A total Positive and Negative Symptoms of Schizophrenia (PANSS) score of >= 60
* A score of >= 16 on Young Mania Rating Scale (YMRS) or a score of >= 16 on the Hamilton Depression Rating Scale (HAM-D 21)

Exclusion Criteria:

* A primary active mental illness diagnosis other than schizoaffective disorder
* Patients with first episode psychosis
* Active substance dependence within previous 6 months
* Treatment with clozapine within 6 months of randomization
* A history of treatment resistance, defined by failure to respond to 2 adequate trials of antipsychotic medication
* Pregnancy, breast-feeding, or planning to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Alphs L, Fu DJ, Turkoz I. Paliperidone for the treatment of schizoaffective disorder. Expert Opin Pharmacother. 2016;17(6):871-83. doi: 10.1517/14656566.2016.1161029. Epub 2016 Mar 24. PMID 26934062
- [Derived] Canuso CM, Lindenmayer JP, Kosik-Gonzalez C, Turkoz I, Carothers J, Bossie CA, Schooler NR. A randomized, double-blind, placebo-controlled study of 2 dose ranges of paliperidone extended-release in the treatment of subjects with schizoaffective disorder. J Clin Psychiatry. 2010 May;71(5):587-98. doi: 10.4088/JCP.09m05564yel. PMID 20492853
- See also: A randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of two dosages of paliperidone ER in the treatment of patients with schizoaffective disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=33&filename=CR010498_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Extended Release (ER) Low Dose: Paliperidone Extended Release (ER) Low Dose - 6mg/day with option to reduce to 3mg/day
- Paliperidone Extended Release (ER) High Dose: Paliperidone Extended Release (ER) High Dose - 12mg/day with option to reduce to 9mg/day
Period: Overall Study
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Started | 107 | 109 | 100
Safety Population: >= 1 Dose of Drug | 107 | 108 | 98
ITT Population | 107 | 105 | 98
Completed | 63 | 72 | 77
Not Completed | 44 | 37 | 23
Not completed — Adverse Event | 7 | 10 | 4
Not completed — Lack of Efficacy | 22 | 12 | 9
Not completed — Lost to Follow-up | 3 | 3 | 3
Not completed — Withdrawal by Subject | 12 | 7 | 5
Not completed — Other | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose | Total
Number analyzed (Participants) | 107 | 105 | 98 | 310
Age Continuous [Mean (Standard Deviation); unit: years] — Intent-to-Treat Population
  years | 37.1 (11.1) | 38.1 (10.0) | 36.5 (10.5) | 37.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-Treat Population
  Participants
    Female | 40 | 35 | 34 | 109
    Male | 67 | 70 | 64 | 201
Region of Enrollment [Number; unit: participants] — Intent-to-Treat Population
  participants
    United States | 39 | 39 | 35 | 113
    India | 33 | 34 | 31 | 98
    Russian Federation | 12 | 13 | 11 | 36
    Ukraine | 23 | 19 | 21 | 63

OUTCOME MEASURES:

1. Primary Outcome: Baseline Positive and Negative Symptoms of Schizophrenia (PANSS) Total Score
Description: The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
Time Frame: Baseline
Population: The Intent-to-Treat population included all randomized participants who received at least 1 dose of study medication (or any portion of a dose) and had both baseline and at least 1 postbaseline PANSS assessment.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a scale | 91.6 (12.5) | 95.9 (13.0) | 92.7 (12.6)

2. Secondary Outcome: Number of Participants With Response
Description: Response is defined as a 30% or more reduction from baseline in PANSS total score and a CGI-C score of <= 2. (CGI-C-SCA: Clinical Global Impression of Change for Schizoaffective Disorder). The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a subject.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population. One patient was not evaluable in the Paliperidone ER Low Dose treatment group.
Measure: Number; unit: count of participants
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 104 | 98
count of participants | 40 | 57 | 62
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; P-value is based on the CMH chi-square test with modified ridit scores, stratified by concomitant medication stratum, and country
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Change in Positive and Negative Symptoms of Schizophrenia (PANSS) Positive Subscale Score
Description: Positive Syndrome Scale (range 7-49): Sum of scores for items 1-7 in positive subscale: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. Higher scores indicate worsening.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: points on subscale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on subscale | -7.9 (6.6) | -9.1 (7.1) | -11.3 (6.3)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p < 0.001, ANCOVA; P-value is from an ANCOVA model with fixed-effects for treatment, concomitant medication stratum, and country, and baseline value as a covariate; LS Means Difference = -3.4, 95% CI [-5.1 to -1.7], Standard Error of Mean 0.9 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.217, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -1.1, 95% CI [-2.8 to 0.6], Standard Error of Mean 0.9 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

4. Secondary Outcome: Change in Positive and Negative Symptoms of Schizophrenia (PANSS) Negative Subscale Score
Description: Negative Syndrome Scale (range 7-49): Sum of scores for items 1-7 in negative subscale: blunted effect, emotional withdrawal, poor rapport, passive apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Higher scores indicate worsening.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: points on a subscale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a subscale | -3.1 (5.1) | -4.4 (5.6) | -4.2 (5.1)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p = 0.108, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Means Difference = -1.0, 95% CI [-2.3 to 0.2], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.430, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -0.5, 95% CI [-1.7 to 0.7], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

5. Secondary Outcome: Change in Positive and Negative Symptoms of Schizophrenia (PANSS) General Psychopathology Subscale Score
Description: General Psychopathology (range 16-112): Sum of scores for somatic concern, anxiety, guilt feelings, tension, mannerisms/posturing, depression, motor retardation, uncooperativeness, unusual thought content, disoriented, poor attention, lack of judgment/insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance. Higher scores indicate worsening.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: points on a subscale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a subscale | -10.7 (11.6) | -13.9 (12.0) | -15.1 (10.3)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p = 0.008, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -3.9, 95% CI [-6.7 to -1.0], Standard Error of Mean 1.5 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.175, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -2.0, 95% CI [-4.8 to 0.9], Standard Error of Mean 1.4 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

6. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Positive Factor Score
Description: Positive PANSS Factor Score (range 8-56): Sum of scores for items 1, 3, 5, and 6 in positive subscale: delusions, hallucinatory behavior, grandiosity, suspiciousness; item 7 in negative subscale: stereotyped thinking; and items 1, 9, and 12 in general psychopathology subscale: somatic concern, unusual thought content, lack of judgment, and insight. Higher scores indicate worsening.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: points on a subscale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a subscale | -6.7 (6.9) | -8.0 (6.8) | -9.6 (6.4)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p = 0.001, ANCOVA; P-value is from an ANCOVA model with fixed-effects for treatment, concomitant medication stratum and country, and baseline value as a covariate; LS Mean Difference = -2.9, 95% CI [-4.6 to -1.1], Standard Error of Mean 0.9 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.209, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -1.1, 95% CI [-2.8 to 0.6], Standard Error of Mean 0.9 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

7. Other Pre Specified Outcome: Hamilton Rating Scale for Depression (HAM-D-21) With Baseline HAM-D-21 Total Score >= 16
Description: Clinician-rated scale that evaluates depressed mood as well as the vegetative and cognitive symptoms of depression. The items are rated on either a 5-point (0 to 4) or a 3-point (0 to 2) scale. The 5-point scale uses a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). Higher scores indicate worsening. The responses are summed to yield the HAM-D-21 score that ranges from 0-63.
Time Frame: Baseline
Population: Intent-to-Treat population with a baseline HAM-D-21 total score of >= 16.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 64 | 76 | 61
points on a scale | 24.4 (5.9) | 25.2 (6.8) | 26.9 (7.3)

8. Other Pre Specified Outcome: Change in Hamilton Rating Scale for Depression (HAM-D-21) With Baseline HAM-D-21 Total Score >= 16
Description: as for outcome 7
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population with a baseline HAM-D-21 total score of >= 16.
Measure: Mean (Standard Deviation); unit: points on scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 64 | 75 | 61
points on scale | -9.9 (10.7) | -13.6 (9.2) | -14.5 (9.2)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p = 0.032, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -3.4, 95% CI [-6.5 to -0.3], Standard Error of Mean 1.6 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.013, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -3.8, 95% CI [-6.8 to -0.8], Standard Error of Mean 1.5 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

9. Secondary Outcome: Change in Positive and Negative Symptoms of Schizophrenia (PANSS) Negative Factor Score
Description: Negative PANSS Factor Score (range 7-49): Sum of scores for items 1, 2, 3, 4, and 6 in negative subscale: blunted affect, emotional withdrawal, poor rapport, passive social withdrawal, lack of spontaneity; and items 7 and 16 in general psychopathology subscale: motor retardation, and active social avoidance. Higher scores indicate worsening.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: points on a subscale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a subscale | -3.0 (5.0) | -4.5 (5.7) | -4.0 (5.1)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p = 0.232, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.7, 95% CI [-2.0 to 0.5], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.310, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.6, 95% CI [-1.8 to 0.6], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

10. Secondary Outcome: Change in Positive and Negative Symptoms of Schizophrenia (PANSS) Disorganized Thought Factor Score
Description: Disorganized Thoughts PANSS Factor Score (range 7-49): Sum of scores for item 2 in positive subscale:Conceptual disorganization; item 5 in negative subscale:difficulty in abstract thinking; and items 5, 10, 11, 13, and 15 in general psychopathology subscale: mannerisms/posturing, disorientation, poor attention, disturbance of volition, and preoccupation. Higher scores indicate worsening.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: points on a subscale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a subscale | -3.7 (5.2) | -5.0 (5.0) | -5.7 (4.8)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p = 0.004, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -1.8, 95% CI [-3.1 to -0.6], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.269, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.7, 95% CI [-1.9 to 0.5], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

11. Secondary Outcome: Change in Positive and Negative Symptoms of Schizophrenia (PANSS) Uncontrolled Hostility/Excitement Factor Score
Description: Uncontrolled Hostility/Excitement PANSS Factor Score (range 4-28): Sum of scores for items 4 and 7 in positive subscale: excitement, hostility; and items 8 and 14 in general psychopathology subscale: uncooperativeness, and poor impulse control. Higher scores indicate worsening.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: points on a subscale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a subscale | -4.8 (4.4) | -5.4 (4.8) | -7.0 (4.2)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -2.1, 95% CI [-3.2 to -1.0], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.314, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.6, 95% CI [-1.7 to 0.5], Standard Error of Mean 0.6 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

12. Secondary Outcome: Change in Positive and Negative Symptoms of Schizophrenia (PANSS) Anxiety/Depression Factor Score
Description: Anxiety/Depression PANSS Factor Score (range 4-28): Sum of scores for items 2, 3, 4, and 6 in general psychopathology subscale: Anxiety, Guilt feelings, Tension, Depression. Higher scores indicate worsening.
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: points on a subscale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a subscale | -3.4 (4.0) | -4.5 (3.8) | -4.3 (3.7)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p = 0.071, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.8, 95% CI [-1.8 to 0.1], Standard Error of Mean 0.5 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.099, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -0.8, 95% CI [-1.7 to 0.1], Standard Error of Mean 0.5 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

13. Secondary Outcome: Clinical Global Impression (CGI-S) - Severity for Schizoaffective Disorder Score at Baseline
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a subject. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill subjects".
Time Frame: Baseline
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on a scale | 4.6 (0.6) | 4.6 (0.6) | 4.6 (0.6)

14. Secondary Outcome: Change in Clinical Global Impression (CGI-S) - Severity for Schizoaffective Disorder
Description: as for outcome 13
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population. One patient was not evaluable in the Paliperidone ER Low Dose treatment group.
Measure: Mean (Standard Deviation); unit: points on scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 104 | 98
points on scale | -1.1 (1.3) | -1.4 (1.2) | -1.8 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Means Difference = -0.6, 95% CI [-0.9 to -0.3], Standard Error of Mean 0.2 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.083, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Means Difference = -0.3, 95% CI [-0.6 to 0.0], Standard Error of Mean 0.2 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

15. Primary Outcome: The Change From Baseline to Week 6 or the Last Post-randomization Assessment During Double-blind Treatment in the Positive and Negative Symptoms of Schizophrenia (PANSS) Total Score.
Description: as for outcome 1
Time Frame: Baseline to Week 6 Last Observation Carried Forward (LOCF) End Point
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: points on scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 105 | 98
points on scale | -21.7 (21.4) | -27.4 (22.1) | -30.6 (19.1)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; One of the primary pairwise comparisons was paliperidone ER high dose vs. placebo. The Hochberg step-up procedure was used to address multiplicity. P-value for between treatment group comparisons is from an ANCOVA model with fixed-effects for treatment, concomitant medication stratum and country, and baseline value as a covariate; Test type: Superiority or Other; p = 0.003, ANCOVA — The Hochberg step-up procedure was used to address multiplicity; [statistical method as in outcome 6, analysis 1]; LS Means Difference = -8.3, 95% CI [-13.8 to -2.9], Standard Error of Mean 2.8 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; One of the primary pairwise comparisons was paliperidone ER low dose vs. placebo. The Hochberg step-up procedure was used to address multiplicity. P-value for between treatment group comparisons is from an ANCOVA model with fixed-effects for treatment, concomitant medication stratum and country, and baseline value as a covariate; Test type: Superiority or Other; p = 0.187, ANCOVA — The Hochberg step-up procedure was used to address multiplicity; [statistical method as in outcome 6, analysis 1]; LS Means Difference = -3.6, 95% CI [-9.0 to 1.8], Standard Error of Mean 2.7 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

16. Secondary Outcome: Clinical Global Impression (CGI-C) - Change for Schizoaffective Disorder
Description: The CGI-C rating scale is a 7 point global assessment that measures the clinician's impression of the change occurring in the illness over a course of treatment, relative to baseline. A rating of 4 is equivalent to "No change". Ratings of <4 are equivalent to "improvement" and ratings of > 4 are equivalent to "worsening".
Time Frame: Week 6 LOCF End Point
Population: Intent-to-Treat population. One patient was not evaluable in the Paliperidone ER Low Dose treatment group.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 107 | 104 | 98
points on a scale | 2.9 (1.4) | 2.6 (1.3) | 2.2 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p < 0.001, ANOVA; P-value is from an ANOVA model with fixed-effects for treatment, concomitant medication stratum and country; LS Means Difference = -0.7, 95% CI [-1.1 to -0.4], Standard Error of Mean 0.2 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher Scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.029, ANOVA; P-value is from an ANOVA model with fixed-effects for treatment, concomitant medication stratum and country; LS Means Difference = -0.4, 95% CI [-0.7 to 0.0], Standard Error of Mean 0.2 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

17. Other Pre Specified Outcome: Young Mania Rating Scale (YMRS) With Baseline YMRS Total Score >= 16
Description: 11-item scale (elevated mood, increased motor activity, sexual interest, sleep, irritability, speech [rate/amount], language-thought disorder, content, disruptive-aggressive behaviors, appearance, and insight) based on subject's report of his or her condition and clinician's behavioral observations during the interview, with emphasis on the latter. Higher scores indicate worsening. The responses are summed to yield the YMRS total score, which ranges from 0 to 60.
Time Frame: Baseline
Population: Intent-to-Treat population with a baseline YMRS total score of >= 16.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 90 | 88 | 79
points on a scale | 28.5 (6.9) | 28.4 (7.4) | 29.9 (8.2)

18. Other Pre Specified Outcome: Change in Young Mania Rating Scale (YMRS) With Baseline YMRS Total Score >= 16
Description: as for outcome 17
Time Frame: Baseline to Week 6 LOCF End Point
Population: Intent-to-Treat population with a baseline YMRS total score of >= 16.
Measure: Mean (Standard Deviation); unit: points on scale
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Number analyzed (Participants) | 90 | 87 | 79
points on scale | -11.5 (11.4) | -14.3 (11.8) | -19.4 (11.7)
Statistical Analysis 1: Comparison: Placebo vs Paliperidone Extended Release (ER) High Dose; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -6.8, 95% CI [-9.9 to -3.7], Standard Error of Mean 1.6 — Paliperidone Extended Release (ER) High Dose - Placebo on the Change Scores. Higher scores indicate worsening
Statistical Analysis 2: Comparison: Placebo vs Paliperidone Extended Release (ER) Low Dose; Test type: Superiority or Other; p = 0.066, ANCOVA; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -2.8, 95% CI [-5.8 to 0.2], Standard Error of Mean 1.5 — Paliperidone Extended Release (ER) Low Dose - Placebo on the Change Scores. Higher scores indicate worsening

ADVERSE EVENTS:
Description: Safety Population
Arm/Group | Placebo | Paliperidone Extended Release (ER) Low Dose | Paliperidone Extended Release (ER) High Dose
Serious Adverse Events (participants affected / at risk) | 6/107 | 10/108 | 2/98
Other Adverse Events (participants affected / at risk) | 61/107 | 78/108 | 68/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=107) | Paliperidone Extended Release (ER) Low Dose (N=108) | Paliperidone Extended Release (ER) High Dose (N=98)
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Salpingitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 2 | 0
Schizoaffective disorder (Psychiatric disorders) | 2 | 4 | 0
Suicidal behavior (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=107) | Paliperidone Extended Release (ER) Low Dose (N=108) | Paliperidone Extended Release (ER) High Dose (N=98)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 5 (8)
Dry Mouth (Gastrointestinal disorders) | 4 (4) | 7 (8) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (9) | 9 (11) | 8 (14)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 5 (5)
Akathisia (Nervous system disorders) | 8 (9) | 4 (4) | 6 (7)
Dizziness (Nervous system disorders) | 7 (7) | 6 (7) | 4 (4)
Headache (Nervous system disorders) | 18 (22) | 15 (16) | 13 (18)
Hypertonia (Nervous system disorders) | 3 (3) | 9 (10) | 4 (5)
Sedation (Nervous system disorders) | 5 (6) | 8 (9) | 4 (5)
Somnolence (Nervous system disorders) | 2 (2) | 5 (5) | 8 (8)
Tremor (Nervous system disorders) | 4 (6) | 13 (13) | 11 (12)
Agitation (Psychiatric disorders) | 6 (6) | 7 (7) | 1 (2)
Insomnia (Psychiatric disorders) | 9 (11) | 5 (6) | 9 (10)
Schizoaffective Disorder (Psychiatric disorders) | 3 (4) | 6 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days